CLINICAL TRIAL: NCT03930771
Title: Capecitabine and Temozolomide for Treatment of Recurrent Pituitary Adenomas
Acronym: TMZ-Cap
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the study had a low accrual rate
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1809019558
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Recurrent Pituitary Adenomas
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Capecitabine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Patients (Experimental): All subjects will receive:
  1. Capecitabine (oral 5-Fluorouracil) 1500mg/m2 orally per day (divided into two doses with maximum daily dose of 2500mg) on days 1 through 14.
  2. Temozolomide (second generation alkylating agent) 150 to 200 mg/m2 orally on days 10 through 14.
  After completion of 6 cycles, patients achieving a complete or partial tumor response may continue to receive capecitabine temozolomide at the investigator's discretion in the absence of disease progression or unacceptable toxicity. Patients will be monitored for six months after they come off the study (either after completing 6 cycles or in setting of disease progression or unacceptable toxicity).
  Interventions: Drug: Capecitabine; Drug: Temozolomide

INTERVENTIONS:
Drug: Capecitabine — 1500mg/m2 orally per day (divided into two doses with maximum daily dose of 2500mg) on days 1 through 14.
Drug: Temozolomide — 150 to 200 mg/m2 orally on days 10 through 14.

SUMMARY:
This is an open label study to assess the efficacy of capecitabine (CAP) and temozolomide (TMZ) in recurrent pituitary adenomas. There will be a safety run-in of at least three patients to establish any dose limiting toxicities. Enrolled patients will receive treatment in 28-day cycles: capecitabine 1500mg/m2 per day (divided into two doses with maximum daily dose of 2500mg) on days 1 through 14 and oral temozolomide 150 to 200 mg/m2 on days 10 through 14. This will be followed by 14 days off treatment. MRI imaging will be completed after every two cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria::

* Male or female ≥ 18 years of age.
* Patients with nonfunctioning tumors must have histologically confirmed pituitary adenoma. Patients with functioning tumors do not require surgery if there is clear diagnosis of functioning pituitary adenomas established based on endocrine evaluation.
* Karnofsky performance status ≥ 70%.
* Life expectancy of greater than six months.
* Residual or recurrent pituitary adenoma ≥1cm in maximal diameter on MRI Brain; patient must have received at least one prior therapy, such as surgery, radiation and/or medical therapy.
* Patients must have normal organ and marrow function as defined below. NOTE: Laboratory values must be taken within 7 days prior to chemotherapy administration. Transfusions and/or growth factor support may not be used to meet this criteria):
* Platelet count ≥ 100 × 109/L.
* Hemoglobin ≥ 9 g/dL.
* WBC ≥ 3 × 109/L
* Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
* Serum bilirubin ≤ 1.5 × upper limit of normal (ULN) or ≤ 3 x ULN if Gilbert's disease is documented.
* Aspartate transaminase (AST) ≤ 2.5 ULN.
* Alanine transaminase (ALT) ≤ 2.5 ULN.
* Serum creatinine ≤ 1.5 × ULN OR creatinine clearance≥60mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Patients must be able to undergo a MRI Brain/Pituitary
* For women of child-bearing potential and for men with partners of child-bearing potential, subject must agree to take contraceptive measures for duration of treatment and at least 6 months after the last dose of chemotherapy.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior temozolomide and/or capecitabine therapy for treatment of the pituitary tumor.
* Other active malignancy outside of nonmelanoma skin cancer (patients in remission and with prior treatment more than two years ago will be accepted into trial).
* Clinically significant renal, hematologic or hepatic abnormalities.
* Use of Vitamin K antagonists such as warfarin (concentrations may be altered by concomitant use of capecitabine)
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics & psychiatric illness/social situations that would limit compliance with study requirements
* History of deficient dihydropyrimidine dehydrogenase activity.
* History of immunodeficiency.
* Patients who are taking any other concurrent investigational therapy.
* Patients who are pregnant or breastfeeding.
* Patients who have had prior radiation treatment in the last six months
* Patients who have had prior pituitary surgery within the last two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Magge, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All subjects will receive:
  1. Capecitabine (oral 5-Fluorouracil) 1500mg/m2 orally per day (divided into two doses with maximum daily dose of 2500mg) on days 1 through 14.
  2. Temozolomide (second generation alkylating agent) 150 to 200 mg/m2 orally on days 10 through 14.
  After completion of 6 cycles, patients achieving a complete or partial tumor response may continue to receive capecitabine temozolomide at the investigator's discretion in the absence of disease progression or unacceptable toxicity. Patients will be monitored for six months after they come off the study (either after completing 6 cycles or in setting of disease progression or unacceptable toxicity).
  Capecitabine: 1500mg/m2 orally per day (divided into two doses with maximum daily dose of 2500mg) on days 1 through 14.
  Temozolomide: 150 to 200 mg/m2 orally on days 10 through 14.
Period: Overall Study
Arm/Group | All Patients
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Radiographic Response, as Defined by the RECIST Criteria.
Description: Evaluation of Target lesions:
  Complete Response (CR):
  Disappearance of all target lesions.
  Partial Response (PR):
  At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD):
  At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum onstudy (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD):
  Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Effect of the CAP and TMZ Combination on Pituitary Function, Measured by Changes in Pituitary Hormone Secretion in Patients
Description: Serum prolactin, IGF-1, ACTH, FSH, LH and TSH levels are used to assess changes in pituitary hormone function. These tests will only be repeated if found to be abnormal at baseline.
Time Frame: At baseline and every 8 weeks, up to 6 months
Measure: Number; unit: ng/mL
Arm/Group | All Patients
Number analyzed (Participants) | 1
ng/mL
  Baseline | 134.7
  Cycle 3 Day 1 | 86.9
  Cycle 5 Day 1 | 69.4
  Cycle 6 Day 1 | 69.8
  End of Treatment | 80.1
  Follow-Up Week 6 | 77.0

3. Secondary Outcome: Safety, as Measured by the Number of Subjects With at Least One AE
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Tolerability of the TMZ and Capecitabine Combination, as Measured by Number of Participants With a Dose-limiting Toxicity
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Tumor Invasiveness and Aggressiveness, Determined by Assessing the Relationship Between Select Indicators With Response to Chemotherapy, Time to Progression, and Tumor Invasiveness.
Description: Tumor invasiveness and aggressiveness, determined by assessing the relationship between select indicators (including Ki67 nuclear labelling index, p53 expression, MGMT expression/methylation status, and additional tumor genetic profiling) with response to chemotherapy, time to progression, and tumor invasiveness (based on the Knosp criteria).
Time Frame: 6 months
Population: Data was not collected in the specified time frame for this outcome measure.
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of consent through six months after completion of the study.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=1)
Fatigue (General disorders) | 1
Paresthesia (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
Due to lower accrual (N=1), there was insufficient data available in order to meet the primary and secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT03930771/Prot_SAP_000.pdf